CLINICAL TRIAL: NCT06730282
Title: A Preliminary Study on the Efficacy of Danggui Shaoyao San and Cuscuta Chinensis in Patients with Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Chia-Ying Chuang, Attending Physician, Department of Chinese Medicine, Taichung Tzu Chi Hospital, Taichung Tzu Chi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC113-20
Record Dates: First submitted 2024-11-24; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-08

CONDITIONS: Primary Dysmenorrhea (PD); Traditional Chinese Medicine (TCM) Approaches
Keywords: Primary Dysmenorrhea; Traditional Chinese Medicine (TCM); Danggui Shaoyao San (DSS); Cuscuta Chinensis (Tu Si Zi); Herbal Medicine
MeSH Terms: interventions — danggui-shaoyao-san; Combined Modality Therapy

STUDY DESIGN:
Intervention Model Description: This study employs a randomized, double-blind, placebo-controlled, parallel assignment model. Participants are randomly allocated to one of four groups: Danggui Shaoyao San (DSS), Cuscuta Chinensis (Tu Si Zi), a combination of DSS and Tu Si Zi, or a placebo group. Each group receives its designated intervention throughout two consecutive menstrual cycles. The parallel design ensures that outcomes can be directly compared between groups without crossover, maintaining the integrity of the treatment effects. The double-blind approach minimizes bias by blinding both participants and investigators to group assignments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this double-blind clinical trial, all participants, care providers, investigators, and outcomes assessors are masked to the group assignments. The study medications (Danggui Shaoyao San, Cuscuta Chinensis, combination therapy, and placebo) are prepared in identical medication containers with no distinguishable labeling. Randomization is conducted using a block randomization scheme, and the allocation sequence is securely managed by the study pharmacy. Neither the study team nor the participants have access to the randomization code until the trial concludes. This ensures unbiased treatment administration and assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Danggui Shaoyao San (Experimental): Participants in this group will receive Danggui Shaoyao San, a traditional Chinese medicine (TCM) formula, for the treatment of primary dysmenorrhea. The medication will be administered starting 3 to 7 days before menstruation and continued until 3 days after menstruation for two consecutive menstrual cycles. Danggui Shaoyao San is intended to regulate blood flow, reduce inflammation, and alleviate uterine contractions associated with dysmenorrhea.
  Interventions: Drug: Danggui Shaoyao San (DSS)
- Cuscuta Chinensis (Experimental): Participants in this group will receive Cuscuta Chinensis, a TCM formula commonly used to support kidney function and alleviate menstrual pain. The medication will be administered starting 3 to 7 days before menstruation and continued until 3 days after menstruation for two consecutive menstrual cycles. This group aims to evaluate the efficacy of Cuscuta Chinensis in managing dysmenorrhea symptoms.
  Interventions: Drug: Cuscuta Chinensis (Tu Si Zi)
- Danggui Shaoyao San + Cuscuta Chinensis (Experimental): articipants in this group will receive a combination of Danggui Shaoyao San and Cuscuta Chinensis. The combined therapy will be administered starting 3 to 7 days before menstruation and continued until 3 days after menstruation for two consecutive menstrual cycles. This group aims to assess whether the combination therapy provides enhanced efficacy in reducing pain and other menstrual symptoms compared to single interventions.
  Interventions: Drug: Combination Therapy (DSS + Tu Si Zi)
- Placebo (Placebo Comparator): Participants in this group will receive a placebo that matches the study medications in appearance and packaging. The placebo will be administered starting 3 to 7 days before menstruation and continued until 3 days after menstruation for two consecutive menstrual cycles. This group serves as a control to evaluate the specific effects of the active interventions on primary dysmenorrhea.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Danggui Shaoyao San (DSS) — Danggui Shaoyao San is a traditional Chinese medicine (TCM) formula used to regulate blood flow, alleviate pain, and reduce inflammation. Participants in this arm will receive DSS starting 3 to 7 days before menstruation and continue until 3 days after menstruation for two cycles.
  Arms: Danggui Shaoyao San
Drug: Cuscuta Chinensis (Tu Si Zi) — Cuscuta Chinensis is a TCM formula traditionally used to nourish kidney essence and improve menstrual health. Participants in this arm will receive Tu Si Zi starting 3 to 7 days before menstruation and continue until 3 days after menstruation for two cycles.
  Arms: Cuscuta Chinensis
Drug: Combination Therapy (DSS + Tu Si Zi) — This intervention combines Danggui Shaoyao San and Cuscuta Chinensis. Participants will receive both formulas starting 3 to 7 days before menstruation and continue until 3 days after menstruation for two cycles.
  Arms: Danggui Shaoyao San + Cuscuta Chinensis
Drug: Placebo — Participants in this arm will receive a placebo that matches the appearance of the study medications. The placebo will be administered on the same schedule as the active treatments for two menstrual cycles.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the efficacy of two traditional Chinese medicine (TCM) formulas, Danggui Shaoyao San (DSS) and Cuscuta Chinensis (Tu Si Zi), in treating primary dysmenorrhea (PD). Primary dysmenorrhea, a common condition characterized by painful menstrual cramps, affects many women of reproductive age and significantly impacts their quality of life. Conventional treatments, such as NSAIDs and oral contraceptives, often have limited efficacy or side effects, underscoring the need for alternative therapeutic options.

In this randomized, double-blind study, participants will be divided into four groups: DSS, Tu Si Zi, a combination of DSS and Tu Si Zi, and a placebo group. The study will measure treatment outcomes using the Visual Analogue Scale (VAS) for pain and the Menstrual Symptom Questionnaire (MSQ), which captures physical and emotional symptoms. Additionally, TCM-based tools like pulse diagnosis and constitution questionnaires will be employed to explore personalized treatment strategies.

This research seeks to determine whether these TCM formulas can alleviate pain and improve other menstrual symptoms, potentially providing broader benefits than conventional painkillers. The findings aim to support evidence-based integration of TCM in managing dysmenorrhea and inform clinicians and patients about effective therapeutic choices.

DETAILED DESCRIPTION:
Study Overview This study investigates the efficacy of two traditional Chinese medicine (TCM) formulations, Danggui Shaoyao San (DSS) and Cuscuta Chinensis (Tu Si Zi), in managing primary dysmenorrhea (PD). PD is a prevalent condition characterized by painful menstrual cramps, often accompanied by physical and emotional symptoms such as fatigue, irritability, nausea, and breast tenderness. Existing treatment options, including NSAIDs and hormonal contraceptives, are effective for symptom relief but may cause side effects or fail to address associated non-pain symptoms, emphasizing the need for complementary or alternative therapies.

Study Design The trial is a randomized, double-blind, placebo-controlled study. Participants meeting the inclusion criteria will be randomly assigned to one of four groups: DSS, Tu Si Zi, a combination of DSS and Tu Si Zi, or placebo. Each treatment will be administered 3 to 7 days prior to menstruation and continued until 3 days post-menstruation. The intervention spans two consecutive menstrual cycles.

The primary outcomes will be changes in pain intensity measured by the Visual Analogue Scale (VAS) and improvements in menstrual symptoms evaluated using the Menstrual Symptom Questionnaire (MSQ). Secondary outcomes include an exploration of the correlation between TCM pulse diagnosis, TCM constitution types, and therapeutic responses, providing insights into the personalization of treatment based on TCM differentiation (辨證).

Rationale Danggui Shaoyao San, a classic TCM formula, is widely used for blood and qi regulation, reducing uterine contractions, and alleviating menstrual pain. Research suggests that it has anti-inflammatory properties and supports immune regulation, making it suitable for patients with blood stasis and qi stagnation patterns. Conversely, Cuscuta Chinensis, traditionally used to nourish kidney essence and yang, may be effective for individuals with kidney deficiency patterns associated with PD. The combination of these formulas could potentially enhance therapeutic outcomes by addressing multiple pathophysiological mechanisms simultaneously.

Methods Eligible participants are women aged 20-45 years with regular menstrual cycles (21-42 days) and a history of moderate to severe menstrual pain (VAS > 3) persisting for at least three cycles. Participants will be excluded if they have secondary dysmenorrhea caused by underlying conditions (e.g., endometriosis), use intrauterine devices, are pregnant or breastfeeding, or are taking anticoagulants or other conflicting medications.

Participants will undergo the following assessments:

Pain and Symptom Evaluation

VAS: Pain intensity will be measured before, during, and after treatment to assess changes.

MSQ: This tool evaluates menstrual symptoms such as mood changes, fatigue, nausea, diarrhea, and abdominal bloating, offering a comprehensive view of symptom burden.

TCM Diagnostic Tools

Pulse Diagnosis: Using a pulse diagnosis device, data from the radial artery will be collected to assess energy distribution across the pulse positions (cun, guan, chi).

TCM Constitution Questionnaire: Participants will complete a validated questionnaire to determine their constitution type, providing context for their treatment response.

Clinical and Demographic Data Collection

Baseline characteristics, including age, BMI, vital signs, and analgesic use, will be recorded.

Blinding and Randomization Randomization will be performed using a block randomization scheme. All participants, investigators, and outcome assessors will be blinded to group assignments. The study medications, prepared in identical capsules, will be indistinguishable from the placebo. The placebo group will serve as a control to isolate the specific effects of the TCM interventions.

Data Analysis The study will use repeated measures ANOVA to evaluate within-group and between-group differences in VAS and MSQ scores over time. Multivariate linear regression will identify variables influencing treatment outcomes, including constitution type and baseline symptom severity. Statistical significance will be set at p < 0.05.

Significance and Expected Outcomes This trial aims to determine whether DSS, Tu Si Zi, or their combination can effectively alleviate menstrual pain and associated symptoms, providing a holistic approach to managing PD. Additionally, it seeks to validate the scientific basis of TCM differentiation in treatment selection, enhancing its integration into modern clinical practice. The findings will inform clinicians and patients about effective, personalized therapeutic options and expand the evidence base for TCM in managing gynecological conditions.

Ethical Considerations The study has been approved by the Institutional Review Board (IRB) of Taichung Tzu Chi Hospital. Participants will provide written informed consent before enrollment. All data will be securely stored and anonymized to protect participant privacy.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged 20 to 45 years.
2. Regular menstrual cycles (21 to 42 days).
3. History of moderate to severe primary dysmenorrhea (Visual Analogue Scale (VAS) score > 3) persisting for at least three consecutive menstrual cycles.
4. Able to understand and complete the study questionnaires (e.g., MSQ).
5. Willing to comply with study protocols, including taking study medications and attending follow-up visits.

Exclusion Criteria:

1. Secondary dysmenorrhea caused by conditions such as endometriosis, pelvic inflammatory disease, or uterine fibroids.
2. Current use of an intrauterine contraceptive device (IUD).
3. Irregular menstrual cycles.
4. Pregnant, breastfeeding, or planning pregnancy within the study period.
5. Use of anticoagulant medications (e.g., aspirin, warfarin, or heparin).
6. Known allergies to any components of the study medications.
7. Severe uncontrolled systemic diseases (e.g., neurological disorders, immunodeficiency, or bleeding disorders).
8. Concurrent use of other herbal medicines or alternative treatments for premenstrual syndrome or dysmenorrhea.
9. Participation in another clinical trial during the study period.

   -

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is open to individuals who self-identify as female and experience menstrual cycles. Eligibility is determined based on biological sex at birth, as the condition being studied, primary dysmenorrhea, specifically affects individuals with a uterus.
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured by the Visual Analogue Scale (VAS) | Baseline and after two menstrual cycles (approximately 8 weeks)
  Pain intensity will be assessed using the Visual Analogue Scale (VAS), where participants rate their pain on a scale of 0 (no pain) to 10 (worst pain imaginable). The change in scores from baseline to post-treatment will be analyzed to evaluate the interventions' effect on reducing primary dysmenorrhea pain.

SECONDARY OUTCOMES:
Change in Menstrual Symptoms Measured by the Menstrual Symptom Questionnaire (MSQ) | Baseline and after two menstrual cycles (approximately 8 weeks)
  The MSQ evaluates physical and emotional menstrual symptoms, such as irritability, fatigue, abdominal pain, nausea, and breast tenderness. Each symptom is rated on a 5-point Likert scale ("Never" to "Always"). Total and individual scores will be analyzed to assess improvements in symptom burden.
Change in the Frequency of Medication Use for Pain Relief | Baseline and after two menstrual cycles (approximately 8 weeks)
  Participants will report the number of times they used pain medication during each menstrual period at baseline and after two menstrual cycles. In addition, the types and doses of pain medications used will be carefully recorded and analyzed to provide a comprehensive evaluation of treatment efficacy.
  For statistical analysis, the mean frequency of medication use will be calculated for each participant at baseline and after two menstrual cycles.
Correlation Between TCM Pulse Diagnosis Parameters and Menstrual Symptom Severity | Baseline and after two menstrual cycles (approximately 8 weeks)
  Radial artery pulse data will be collected using a TCM pulse diagnosis device, which measures parameters across three positions: cun, guan, and chi on both the left and right wrists. Each position's waveforms will be analyzed within frequency bands of 0-10Hz, 10-50Hz, and 13-50Hz. Additional parameters, such as SER and EP waveforms, represent distinct characteristics of the radial artery pulse.
  Pulse data will be correlated with symptom severity, as assessed by the Menstrual Symptom Questionnaire (MSQ), to identify patterns or relationships. This analysis aims to explore how pulse energy distributions and waveform variations reflect changes in symptom intensity and treatment outcomes.
Correlation Between TCM Constitution and Treatment Outcomes Using the Body Constitution Questionnaire (BCQ) | Baseline and after two menstrual cycles (approximately 8 weeks)
  The Body Constitution Questionnaire (BCQ) will be used to assess participants' TCM constitution types, including Yang-deficiency, Yin-deficiency, and Stasis. Participants will rate 44 items on a 5-point scale, reflecting the frequency or severity of symptoms over the past month. The study will analyze correlations between changes in BCQ constitution scores and treatment outcomes, including improvements in pain intensity (VAS) and menstrual symptoms (MSQ), to explore the role of TCM constitution in predicting therapeutic efficacy.

OTHER OUTCOMES:
Change in Non-Pain Symptoms of Menstruation | Baseline and after two menstrual cycles (approximately 8 weeks)
  Non-pain symptoms of menstruation will be assessed using specific items from the Menstrual Symptom Questionnaire (MSQ), including abdominal bloating, nausea, irritability, anxiety, and fatigue. Each symptom is rated on a 5-point Likert scale ranging from "Never" to "Always."
  For statistical analysis, the mean scores of individual non-pain symptom items will be calculated for each participant at baseline and after two menstrual cycles.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Tzu Chi Hospital, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study will be made available to researchers upon reasonable request. The shared data will include all primary and secondary outcome measures as defined in the protocol, along with de-identified demographic and clinical information. Supporting documents, such as the study protocol, statistical analysis plan, and informed consent form, will also be shared to ensure transparency and reproducibility of results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start Date: Data will be available 6 months after the publication of primary results.
  End Date: Data will remain accessible for up to 5 years following publication.
Access Criteria: Researchers seeking access must submit a written request to the study director, Chung Chia Ying, at jiainwhh@tzuchi.com.tw. Requests must include a detailed research proposal that specifies the intended use of the data and has received approval from an independent ethics review board. Access to the data will require signing a data use agreement, which includes terms to ensure the data are used solely for the proposed purposes and maintained confidentially.